CLINICAL TRIAL: NCT00909974
Title: Effect of Prenatal Nutritional Supplementation on Birth Outcome in Hounde District, Burkina Faso
Acronym: MISAME2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University Ghent (Other); Flemish Interuniversity Council (VLIR) (Network); Nutrition Third World, Belgium (Other)
Responsible Party: Prof. Patrick Kolsteren, head of Child Health and Nutrition Unit, Institute of Tropical Medicine, Belgium
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZEIN2004PR298
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Intrauterine Growth Retardation; Low Birth Weight
Keywords: multiple micronutrients; energy deficiency
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Food supplement (FS) (Experimental): Recipe of food supplement: 33% peanut butter, 32% soy flour, 15% vegetable oil, 20% sugar, UNIMMAP in powdered form Nutritional composition (per dose of 72g) Energy 1.56 MJ, protein 14.7 g, vitamin A 881 µg, vitamin E 13 mg, vitamin D 5 µg, vitamin B1 1.4 mg, vitamin B2 1.4 mg, niacin 21 mg, vitamin B6 1.9 mg, vitamin B12 2.6 µg, folic acid 461 µg, vitamin C 70 mg, iron 30 mg, zinc 15 mg, copper 2 mg, selenium 65 µg, and iodine 150 µg
  Interventions: Dietary Supplement: Food supplement enriched with multiple micronutrients
- UNIMMAP (Active Comparator): UNIMMAPin tablet form: vitamin A 800µg, vitamin E 10 mg, vitamin D 5 µg, vitamin B1 1.4 mg, vitamin B2 1.4 mg, niacin 18 mg, vitamin B6 1.9 mg, vitamin B12 2.6 µg, folic acid 400 µg, vitamin C 70 mg, iron 30 mg, zinc 15 mg, copper 2 mg, selenium 65 µg, and iodine 150 µg
  Interventions: Dietary Supplement: UNIMMAP - multiple micronutrients

INTERVENTIONS:
Dietary Supplement: UNIMMAP - multiple micronutrients — Daily supplementation of one UNIMMAP tablet
  multiple micronutrient supplements (MMN): UNIMMAP: vitamin A 800µg, vitamin E 10 mg, vitamin D 5 µg, vitamin B1 1.4 mg, vitamin B2 1.4 mg, niacin 18 mg, vitamin B6 1.9 mg, vitamin B12 2.6 µg, folic acid 400 µg, vitamin C 70 mg, iron 30 mg, zinc 15 mg, copper 2 mg, selenium 65 µg, and iodine 150 µg
  Arms: UNIMMAP
Dietary Supplement: Food supplement enriched with multiple micronutrients — One dose of 72g per day during whole pregnancy
  Recipe of food supplement: 33% peanut butter, 32% soy flour, 15% vegetable oil, 20% sugar, UNIMMAP in powdered form Nutritional composition (per dose of 72g) Energy 1.56 MJ, protein 14.7 g, vitamin A 881 µg, vitamin E 13 mg, vitamin D 5 µg, vitamin B1 1.4 mg, vitamin B2 1.4 mg, niacin 21 mg, vitamin B6 1.9 mg, vitamin B12 2.6 µg, folic acid 461 µg, vitamin C 70 mg, iron 30 mg, zinc 15 mg, copper 2 mg, selenium 65 µg, and iodine 150 µg
  Other Names: Lipid based nutritional supplement (LNS)
  Arms: Food supplement (FS)

SUMMARY:
Low birth weight (LBW; birth weight<2,500g) is the most important determinant of mortality and morbidity in the neonatal period. It is also a very important factor in predicting nutritional status, health and development in childhood. It even influences health in adult life, contributing to the vicious cycle of disease and poverty. The high rate LBW in DCs represents therefore a major public health problem. Maternal chronic energy deficiency is assumed to be a major determinant of the problem in these countries along with prenatal micronutrient deficiencies. A large body of recent evidence points out that multiple micronutrient supplementation as such has only a modest beneficial effect on fetal growth. Therefore, it is expected that providing these multiple micronutrients in a food supplement covering energy requirement needs of pregnant women will have an effect of public health importance on children's health.

This study has the objective of improving children's health by improving birth outcome and fetal growth through the provision of a food supplement enriched in multimicronutrients during pregnancy.

This research includes 2 constituents:

1. a pilot phase during which dietary behavior of pregnant women is assessed as a component for optimal fetal growth
2. a randomized, placebo-controlled trial, including 1300 pregnant women aimed at testing 2 hypotheses: supplementing pregnant women with a food supplement containing a multivitamin-minerals mix will improve fetal growth; improved fetal growth will have a positive effect on health and growth during infancy.

The trial is planned in Hounde District, Burkina Faso, in collaboration with Centre Muraz, which plays a leader role in research and services providing at the district level and in policy recommendations at the national level. This will ensure that the study findings are incorporated into on-going district programs with possible replication at the national level. The research lasts from February 2006 to August 2009.

DETAILED DESCRIPTION:
Low birth weight (LBW; birth weight<2500g) is an important predictor of mortality and morbidity in the neonatal period of early postnatal growth and growth during childhood. It is also associated with cognitive and behavioral development in the first years of life, health status during childhood, and adult health and human capital. As much as 16 % of all live births worldwide present a LBW, more than 90% being in low-income countries. Rates are particularly high in Asia and sub-Saharan countries. In Burkina Faso, it is estimated that 19 % of all live births in 1999-2005 were LBW.

In developing countries, most cases of LBW are attributed to intrauterine growth retardation (IUGR) rather than to preterm delivery. Factors interacting with fetal development are numerous. Among them maternal malnutrition, particularly energy and micronutrient deficiencies, and malaria during pregnancy are assumed to be major determinants of IUGR. Dietary surveys have consistently shown that multiple micronutrient deficiencies, rather than single deficiencies, are common. However, a number of randomized clinical trials in various countries have shown only a modest beneficial effect on fetal growth when providing multiple micronutrient supplements during pregnancy compared to folic acid and iron supplementation. It is expected that chronic energy deficiency during pregnancy could be hampering the full potential of the effect of multiple micronutrient supplementation. Therefore it is expected that incorporating multiple micronutrients in a food supplement (FS), that provides supplementary energy and protein, instead of multiple micronutrients (UNIMMAP), could have an effect of public health importance on fetal growth and its correlates. The UNIMMAP supplement composition, incorporated in the FS or given in the form of a tablet, was proposed by an expert committee organized by UNICEF, WHO and UNU for pregnancy and lactating women.

The study takes place in the health district of Houndé (south-west of Burkina Faso) in the surroundings of 2 health centers (12,000 inhabitants) from June 2003 to October 2006. Houndé is situated in a Sudano-Sahelian climate belt. The diet is essentially cereal-based. In 2004 and 2006, food consumption surveys estimated the average caloric intake during pregnancy at 8.6 MJ and 8.1 MJ during the postharvest and pre-harvest season respectively. Malaria transmission is permanent with seasonal variations. In 2002, the HIV prevalence among consulting pregnant women in the district was estimated at 2 %. The incidence of LBW in term infants was around 17% at the District Hospital in 2000-2001.

The recruitment of participants is community-based. During a preliminary census, houses in the study area are mapped and numbered and a unique identification code allocated to every woman of child-bearing age. Thirty locally trained home-visitors visit monthly every compound for early detection of pregnancy and referral to the health center for pregnancy test. Once the pregnancy is confirmed and after extensive explanation of the study purposes and procedures in Bwamu, Moré or Dioula, participants are asked to provide signed consent or thumbprints. There are no exclusion criteria other than planning to leave the area within the next 2 years.

This study is a randomized controlled trial, with directly observed supplement intake. Pregnant women are randomly assigned to receive daily either UNIMMAP tablet ( vitamin A 800µg, vitamin E 10 mg, vitamin D 5 µg, vitamin B1 1.4 mg, vitamin B2 1.4 mg, niacin 18 mg, vitamin B6 1.9 mg, vitamin B12 2.6 µg, folic acid 400 µg, vitamin C 70 mg, iron 30 mg, zinc 15 mg, copper 2 mg, selenium 65 µg, and iodine 150 µg) until delivery, or either a food supplement containing the UNIMMAP. The food supplement consists of 33% peanut butter, 32% heat-treated soy flour, 15% vegetable oil, 20% plain sugar and the UNIMMAP micronutrient cocktail in powdered form. Each participant allocated to the FS study group will receive 72g of FS daily which provides 1.56 MJ (372 kcal) of energy and 14.7g protein. The supplement is produced by a local women's association in collaboration with a food technologist, the micronutrients in the FS are dosed by a laboratory technician. UNIMMAP micronutrient tablets are manufactured by Scanpharm (Copenhagen, Denmark). A randomization scheme is generated by a computer program in permuted blocks of 4. Randomization numbers are sealed in opaque envelopes by administrative staff. At each inclusion, the consulting physician in the field opens the next sealed envelope and transmits the randomization number in case of MMN to a pharmacist managing for the packaging of drugs in individual plastic zip sachets containing 31 tablets. In case the randomization number shows allocation to the FS group, the responsible of the FS production site together with project staff, prepares a plastic bag containing 31 FS sachets.

Participants are also randomly assigned randomized to receive intermittent malaria prophylaxis by either two doses or more than two doses of combined sulfadoxine-pyrimethamine (a single dose represented 1500 mg sulfadoxine and 75mg pyrimethamine). The malaria component will be analysed separately.

In case of maternal illness, appropriate treatments are provided according to national guidelines. Severely anemic women (hemoglobin < 70 g/L, without dyspnea) receive ferrous sulphate (200 mg) + folic acid (0.25 mg) twice daily, during 3 months whatever their allocation group. All participants also receive Albendazole 400 mg in the second and third trimester. In case of malaria episode despite the preventative treatment, quinine (300 mg, 3 times a day) is given during 5 days. Vitamin A (200.000 IU) is given to all women after delivery, in conformity with the national recommendations.

ELIGIBILITY:
Inclusion Criteria:

* All the women of child-bearing age (15-44 years) living in the study area (4 100) will be visited monthly to assess early pregnancy and will be invited to participate in the trial.

Exclusion Criteria:

* planning to move outside the district within the 2 years following the start of the trial.
* regularly using a contraceptive method.
* already pregnant at the start of the trial.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1302 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Weight, length and Rohrer index at birth, and gestational duration in singleton pregnancies. | At birth
Mortality, morbidity and growth during the first year of life | Monthly during infancy

SECONDARY OUTCOMES:
Placental weight; LBW; SGA; thoracic circumference; head circumference; mid-upper arm circumference; hemoglobin concentration in mothers and in newborns; soluble sTfR in cord blood as an iron status indicator; preterm birth; stillbirth; perinatal death | Different depending on mother and child

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Huybregts, MSc, Principal Investigator — University Ghent, Belgium; Patrick Kolsteren, PhD, Study Chair — Institute of Tropical Medicine, Belgium; Ghent University, Belgium; Dominqiue Roberfroid, MD, Principal Investigator — Institute of Tropical Medicine, Belgium; Nicolas Meda, PhD, Principal Investigator — Centre Muraz
Locations (1):
- Centre Muraz, 2054, Avenue Mamadou KONATE, Bobo-Dioulasso, Burkina Faso

REFERENCES:
- [Derived] Toe LC, Bouckaert KP, De Beuf K, Roberfroid D, Meda N, Thas O, Van Camp J, Kolsteren PW, Huybregts LF. Seasonality modifies the effect of a lipid-based nutrient supplement for pregnant rural women on birth length. J Nutr. 2015 Mar;145(3):634-9. doi: 10.3945/jn.114.203448. Epub 2015 Jan 14. PMID 25733482
- [Derived] Lanou H, Huybregts L, Roberfroid D, Nikiema L, Kouanda S, Van Camp J, Kolsteren P. Prenatal nutrient supplementation and postnatal growth in a developing nation: an RCT. Pediatrics. 2014 Apr;133(4):e1001-8. doi: 10.1542/peds.2013-2850. Epub 2014 Mar 3. PMID 24590752
- [Derived] Huybregts L, Roberfroid D, Lanou H, Meda N, Taes Y, Valea I, D'Alessandro U, Kolsteren P, Van Camp J. Prenatal lipid-based nutrient supplements increase cord leptin concentration in pregnant women from rural Burkina Faso. J Nutr. 2013 May;143(5):576-83. doi: 10.3945/jn.112.171181. Epub 2013 Mar 27. PMID 23535609
- [Derived] Valea I, Tinto H, Drabo MK, Huybregts L, Sorgho H, Ouedraogo JB, Guiguemde RT, van Geertruyden JP, Kolsteren P, D'Alessandro U; FSP/MISAME study Group. An analysis of timing and frequency of malaria infection during pregnancy in relation to the risk of low birth weight, anaemia and perinatal mortality in Burkina Faso. Malar J. 2012 Mar 16;11:71. doi: 10.1186/1475-2875-11-71. PMID 22433778
- [Derived] Huybregts L, Roberfroid D, Lanou H, Menten J, Meda N, Van Camp J, Kolsteren P. Prenatal food supplementation fortified with multiple micronutrients increases birth length: a randomized controlled trial in rural Burkina Faso. Am J Clin Nutr. 2009 Dec;90(6):1593-600. doi: 10.3945/ajcn.2009.28253. Epub 2009 Oct 7. PMID 19812173
- See also: Institute of Tropical Medicine Prince Leopold, Antwerp, Belgium — http://www.itg.be